CLINICAL TRIAL: NCT01925976
Title: Individualized Tailor-made Dietetic Intervention Program at Schools Enhances Eating Behaviors and Dietary Habits in Obese Hispanic Children of Low Socioeconomic Status
Brief Title: Individualized Dietetic Intervention-eating Habits in Obese Hispanic Children of Low Socioeconomic Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Tecnologico y de Estudios Superiores de Monterey (Other)
Responsible Party: Principal Investigator, Leticia Elizondo-Montemayor, M.D., Instituto Tecnologico y de Estudios Superiores de Monterey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIETARYHABITS2012-CINCO
Record Dates: First submitted 2013-08-14; First posted 2013-08-20 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Overweight; Obesity
Keywords: obesity; dietetic intervention; eating behaviors; children; healthy eating; energy dense foods
MeSH Terms: conditions — Overweight; Obesity; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Individualized dietetic intervention (Other): Behavioral: Individualized dietetic intervention-eating habits.
  Interventions: Behavioral: Individualized dietetic intervention-eating habits

INTERVENTIONS:
Behavioral: Individualized dietetic intervention-eating habits — The school-year (12 months) dietetic intervention consisted of anthropometric measurements, dietetic assessment, energy restriction tailor-made daily menus, and parental education every three weeks at each school site.
  Other Names: tailor-made dietetic intervention

SUMMARY:
The purpose of this study is to implement an individualized, face-to-face, parent supported and school-partnership dietetic intervention program to promote healthy eating habits in obese, Hispanic, children from low socioeconomic status due to the high predisposition to unhealthy eating habits and obesity in this population.

DETAILED DESCRIPTION:
Study Population An open invitation is made to children from eight public schools of low socioeconomic status (low SES), representative of all geographical areas of Monterrey, second largest city in México. From those that accept, children will be randomly selected and screened for overweight/obesity using BMI percentiles, and those who qualify for overweight/obesity will be invited to participate in the dietetic intervention program.

Clinical Evaluation Based on the World Health Organization and the American Academy of Pediatrics criteria (BA, Spear, et al., 2007), overweight is considered as BMI > 85th and < 95th percentiles and obesity as > 95th percentile according to age and sex. Anthropometric measurements will be performed in all participants at each school. Standing height will be determined to the nearest 0.5 cm (portable Seca® stadiometer, North America) and weight to the nearest 0.1 kg while children wear light clothing, no socks or shoes (TANITA TBF 300® scale, Arlington, Illinois). Waist circumference will be measured to the nearest 0.1 cm at the level of the umbilicus with a flexible fiberglass tape while the subjects are standing, after gently exhaling, and with no clothing on the area. BMI will be calculated by weight (kg) divided by the square of height (m). Measurements will be performed by the same three trained registered dietitians (RD) in all children to control the inter-observer variability.

Dietetic Intervention The principal strategies for the change in energy and food groups consumption, are dietary modifications for the children and parental support, as recommended by national associations (SR, Daniels et al, 2009; TA, Nicklas, et al, 2008; BA, Spear, et al., 2007, A Report of the Panel on Macronutrients et al, 2005). Dietetic intervention will be given individually by a RD for every child at each school, every three weeks, for a total of 13 visits during the school-year. Children will leave the classroom to attend the 30-minute nutrition counseling. Each child will be seen by the same RD throughout the school-year to favor compliance to the plan and to avoid inter-examiner bias. Each session will consist of: 1.) Anthropometric assessment; 2.) Dietetic assessment by means of 24-hour diet recalls, a standardized food frequency questionnaire that included Mexican foods, and food replicas to aid in estimation of portion sizes; 3.) Individualized energy restriction and balanced macronutrient dietary planning; 4.) Provision of structured, tailored-made daily menus and meals for the next three weeks for each child; and 5.) Information given to parents/care givers about healthy food, eating practices and portion sizes. Attendance of the parent/care giver is mandatory to help answer the 24-hour recalls and to assure commitment to follow the dietary recommendations at home. After each visit, the RD will record the information into the software (NutriKcal®VO software, Consinfo S.C., D.F., Mexico.), which determines energy intake and diet composition.

Diet composition (macronutrients) is based on the most recent dietary recommended intake for children (A Report of the Panel on Macronutrients et al, 2005) : 25%-35% of total calories from fat; 45%-65% from carbohydrates and 10%-30% from protein. Additional recommendations for children or adolescents include a variety of foods low in saturated fat (<10% kcal), no trans fat and cholesterol <300 mg/day. The RDs will promote age appropriate serving sizes, including approximately >5 servings of fruit and vegetables, >3 servings of low fat milk or dairy products, >6 servings of whole-grain products per day; increase of dietary fiber and reduction of salt intake (US Department of Agriculture and US Department of Health and Human Services, 2010). As well, children will be advised to avoid overconsumption of energy dense, nutrient-poor foods and beverages (TA, Nicklas et al, 2008).

Reduction in calorie intake is approached following the recommendations of the American Heart Association in which children > 4 years old with a BMI > 85th percentile to achieve BMI percentile reductions to <85th percentile with weight maintenance during linear growth (SR, Daniels, et al, 2009). As advised (BA, Spear, et al, 2007), progressive restriction of 150-900 calories from actual intake throughout the school year is recommended so that obese children with BMI >95th percentile lose gradually 0.5 kilogram/month and those with BMI >99th percentile lose a maximum of 0.9 kilogram/week.

Statistical Methods MINITAB version 16 (Minitab Inc., State College, Pennsylvania, USA) will be used to analyze the differences between anthropometric parameters and nutrient intake values at baseline and end of intervention; Microsoft Excel 2007 (Microsoft Corp., Redmond, Washington, USA) will be used to incorporate the input of data. The results will be expressed as mean ± standard deviation (s.d.) and their corresponding 95% confidence intervals (CI). Comparisons between groups for dependent variables will be made using paired Student's t-test for means. The mean comparisons between gender groups will be determined using t-test for independent samples. All tests will be interpreted based on two-tailed hypothesis. The significance level will be set at 0.05 in all cases.

ELIGIBILITY:
Inclusion Criteria:

* Attendance from first to sixth grade
* Ages 6-12 years
* BMI ≥ 85th percentile for age and sex
* Hispanic origin
* Both parents Hispanic
* Low socioeconomic status
* Signed consent from both parents/care givers and active assent from children

Exclusion Criteria:

* Disapproval by the children's physician due to any at-risk medical condition known by the parents

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in energy dense food consumption at 12 months | 12 months
  Energy dense food will include: processed meats, oils, saturated fat, sweets, sweetened beverages, desserts, refined-grain bakery, sweets, chips, fries, whole-fat milk, and fast foods. Measured in servings per day and servings per week. Results will be expressed in mean ± standard deviation for each and their corresponding 95% confidence intervals for the mean difference at baseline and 12 months.
Change from baseline in nutrient dense food consumption at 12 months | 12 months
  Nutrient dense food will include: fruits, vegetables, whole grains, beans and peas, fish/poultry. Measured in servings per day and servings per week. Results will be expressed in mean ± standard deviation for each and their corresponding 95% confidence intervals for the mean difference at baseline and 12 months.

SECONDARY OUTCOMES:
Change from baseline in waist circumference at 12 months | 12 months
  Waist circumference measured in centimeters. The results will be expressed as mean ± standard deviation and its corresponding 95% confidence intervals for the mean difference at baseline and 12 months.
Change from baseline in total energy intake at 12 months | 12 months
  Energy intake assessed according to a 24-hour food recall and reported in kilocalories per day. The results will be expressed as mean ± standard deviation and its corresponding 95% confidence intervals for the mean difference at baseline and 12 months.
Change from baseline in carbohydrate consumption at 12 months | 12 months
  Carbohydrate consumption will be expressed as energy intake in kilocalories per day, quantity in grams and percent of calories from the diet. The results will be expressed as mean ± standard deviation for each and their corresponding 95% confidence intervals for the mean difference at baseline and 12 months.
Change from baseline in protein consumption at 12 months | 12 months
  Protein consumption will be expressed as energy intake in kilocalories per day, quantity in grams and percent of calories from the diet. The results will be expressed as mean ± standard deviation for each and their corresponding 95% confidence intervals for the mean difference at baseline and 12 months.
Change from baseline in fat consumption at 12 months | 12 months
  Fat consumption will be expressed as energy intake in kilocalories per day, quantity in grams and percent of calories from the diet. The results will be expressed as mean ± standard deviation for each and their corresponding 95% confidence intervals for the mean difference at baseline and 12 months.
Change from baseline in water consumption at 12 months | 12 months
  Water consumption will be expressed as a mean ± standard deviation and its corresponding 95% confidence intervals for the mean difference at baseline and 12 months.
Change from baseline in body mass index percentile at 12 months | 12 months
  Body mass index (BMI) calculated by weight in kilograms (kg) divided by the square of height in meters (m). Measurements at baseline and 12 months. Results will be reported for BMI percentile according to the Body mass index-for-age percentiles: 2 to 20 years for boys and girls respectively, from the Centers for Disease and Control Prevention (CDC) Growth Charts: United States (http://www.cdc.gov/growthcharts). The results will be expressed as mean ± standard deviation and their corresponding 95% confidence intervals for the mean difference at baseline and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Leticia Elizondo-Montemayor, M.D., Principal Investigator — Instituto Tecnologico y de Estudios Superiores de Monterrey
Locations (1):
- Clinical Nutrition and Obesity Research Center. School of Medicine and Health Sciences, TEC Salud, Tecnológico de Monterrey, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Daniels SR, Jacobson MS, McCrindle BW, Eckel RH, Sanner BM. American Heart Association Childhood Obesity Research Summit Report. Circulation. 2009 Apr 21;119(15):e489-517. doi: 10.1161/CIRCULATIONAHA.109.192216. Epub 2009 Mar 30. No abstract available. PMID 19332458
- [Background] Secretaría de Salud. México avanza en la cobertura universal de salud: Felipe Calderón. México Sano. 2009;8:3
- [Background] Olaiz-Fernández G, Rivera-Dommarco J, Shamah-Levy T, et al. Encuesta Nacional de Salud y Nutrición 2012: resultados nacionales [Internet]. Cuernavaca, México: Instituto Nacional de Salud Pública (MX) 2012 [cited 2012 July]. 200p. Available from: http://ensanut.insp.mx/informes/ENSANUT2012ResultadosNacionales.pdf
- [Background] Elizondo-Montemayor L, Serrano-Gonzalez M, Ugalde-Casas PA, Cuello-Garcia C, Borbolla-Escoboza JR. Metabolic syndrome risk factors among a sample of overweight and obese Mexican children. J Clin Hypertens (Greenwich). 2010 May;12(5):380-7. doi: 10.1111/j.1751-7176.2010.00263.x. PMID 20546382
- [Background] Cook S, Weitzman M, Auinger P, Nguyen M, Dietz WH. Prevalence of a metabolic syndrome phenotype in adolescents: findings from the third National Health and Nutrition Examination Survey, 1988-1994. Arch Pediatr Adolesc Med. 2003 Aug;157(8):821-7. doi: 10.1001/archpedi.157.8.821. PMID 12912790
- [Background] Fuentes-Afflick E, Hessol NA. Overweight in young Latino children. Arch Med Res. 2008 Jul;39(5):511-8. doi: 10.1016/j.arcmed.2008.02.008. Epub 2008 Apr 8. PMID 18514096
- [Background] Mazur RE, Marquis GS, Jensen HH. Diet and food insufficiency among Hispanic youths: acculturation and socioeconomic factors in the third National Health and Nutrition Examination Survey. Am J Clin Nutr. 2003 Dec;78(6):1120-7. doi: 10.1093/ajcn/78.6.1120. PMID 14668273
- [Background] Rodriguez-Ramirez S, Mundo-Rosas V, Garcia-Guerra A, Shamah-Levy T. Dietary patterns are associated with overweight and obesity in Mexican school-age children. Arch Latinoam Nutr. 2011 Sep;61(3):270-8. PMID 22696895
- [Background] Eagle TF, Sheetz A, Gurm R, Woodward AC, Kline-Rogers E, Leibowitz R, Durussel-Weston J, Palma-Davis L, Aaronson S, Fitzgerald CM, Mitchell LR, Rogers B, Bruenger P, Skala KA, Goldberg C, Jackson EA, Erickson SR, Eagle KA. Understanding childhood obesity in America: linkages between household income, community resources, and children's behaviors. Am Heart J. 2012 May;163(5):836-43. doi: 10.1016/j.ahj.2012.02.025. PMID 22607862
- [Background] Wang Y, Beydoun MA. The obesity epidemic in the United States--gender, age, socioeconomic, racial/ethnic, and geographic characteristics: a systematic review and meta-regression analysis. Epidemiol Rev. 2007;29:6-28. doi: 10.1093/epirev/mxm007. Epub 2007 May 17. PMID 17510091
- [Background] Kendzor DE, Caughy MO, Owen MT. Family income trajectory during childhood is associated with adiposity in adolescence: a latent class growth analysis. BMC Public Health. 2012 Aug 5;12:611. doi: 10.1186/1471-2458-12-611. PMID 22863369
- [Background] Ogden CL, Lamb MM, Carroll MD, Flegal KM. Obesity and socioeconomic status in children and adolescents: United States, 2005-2008. NCHS Data Brief. 2010 Dec;(51):1-8. PMID 21211166
- [Background] Nicklas TA, Hayes D; American Dietetic Association. Position of the American Dietetic Association: nutrition guidance for healthy children ages 2 to 11 years. J Am Diet Assoc. 2008 Jun;108(6):1038-44, 1046-7. doi: 10.1016/j.jada.2008.04.005. PMID 18564454
- [Background] Spear BA, Barlow SE, Ervin C, Ludwig DS, Saelens BE, Schetzina KE, Taveras EM. Recommendations for treatment of child and adolescent overweight and obesity. Pediatrics. 2007 Dec;120 Suppl 4:S254-88. doi: 10.1542/peds.2007-2329F. PMID 18055654
- [Background] Vereecken C, Legiest E, De Bourdeaudhuij I, Maes L. Associations between general parenting styles and specific food-related parenting practices and children's food consumption. Am J Health Promot. 2009 Mar-Apr;23(4):233-40. doi: 10.4278/ajhp.07061355. PMID 19288844
- [Background] Mendoza JA, Watson K, Cullen KW. Change in dietary energy density after implementation of the Texas Public School Nutrition Policy. J Am Diet Assoc. 2010 Mar;110(3):434-40. doi: 10.1016/j.jada.2009.11.021. PMID 20184994
- [Background] Katz DL, O'Connell M, Njike VY, Yeh MC, Nawaz H. Strategies for the prevention and control of obesity in the school setting: systematic review and meta-analysis. Int J Obes (Lond). 2008 Dec;32(12):1780-9. doi: 10.1038/ijo.2008.158. PMID 19079319
- [Background] Muller MJ, Danielzik S, Pust S. School- and family-based interventions to prevent overweight in children. Proc Nutr Soc. 2005 May;64(2):249-54. doi: 10.1079/pns2005424. PMID 15960869
- [Background] A Report of the Panel on Macronutrients, Subcommittees on Upper Reference Levels of Nutrients and Interpretation and Uses of Dietary Reference Intakes, and the Standing Committee on the Scientific Evaluation of Dietary Reference Intakes; Food and Nutrition Board; and Institute or Medicine. Dietary Reference Intakes for Energy, Carbohydrate, Fiber, Fat, Fatty Acids, Cholesterol, Protein, and Amino Acids. Washington, DC: The National Academies Press [Internet]. United States: The National Academies Press, 2005 [cited 2012 July]. 1357 p. Available from: http://www.nap.edu/openbook.php?isbn=0309085373
- [Background] McGuire S. U.S. Department of Agriculture and U.S. Department of Health and Human Services, Dietary Guidelines for Americans, 2010. 7th Edition, Washington, DC: U.S. Government Printing Office, January 2011. Adv Nutr. 2011 May;2(3):293-4. doi: 10.3945/an.111.000430. Epub 2011 Apr 30. No abstract available. PMID 22332062
- [Background] Lioret S, Touvier M, Lafay L, Volatier JL, Maire B. Dietary and physical activity patterns in French children are related to overweight and socioeconomic status. J Nutr. 2008 Jan;138(1):101-7. doi: 10.1093/jn/138.1.101. PMID 18156411
- [Background] McCaffrey TA, Rennie KL, Kerr MA, Wallace JM, Hannon-Fletcher MP, Coward WA, Jebb SA, Livingstone MB. Energy density of the diet and change in body fatness from childhood to adolescence; is there a relation? Am J Clin Nutr. 2008 May;87(5):1230-7. doi: 10.1093/ajcn/87.5.1230. PMID 18469244
- [Background] Newby PK, Muller D, Hallfrisch J, Qiao N, Andres R, Tucker KL. Dietary patterns and changes in body mass index and waist circumference in adults. Am J Clin Nutr. 2003 Jun;77(6):1417-25. doi: 10.1093/ajcn/77.6.1417. PMID 12791618
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Rolls BJ, Drewnowski A, Ledikwe JH. Changing the energy density of the diet as a strategy for weight management. J Am Diet Assoc. 2005 May;105(5 Suppl 1):S98-103. doi: 10.1016/j.jada.2005.02.033. PMID 15867904
- [Background] Senese LC, Almeida ND, Fath AK, Smith BT, Loucks EB. Associations between childhood socioeconomic position and adulthood obesity. Epidemiol Rev. 2009;31:21-51. doi: 10.1093/epirev/mxp006. Epub 2009 Jul 31. PMID 19648176
- [Background] Jackson EA, Eagle T, Leidal A, Gurm R, Smolarski J, Goldberg C, Rogers B, Eagle KA. Childhood obesity: A comparison of health habits of middle-school students from two communities. Clin Epidemiol. 2009 Aug 9;1:133-9. doi: 10.2147/clep.s7609. PMID 20865095
- [Background] Thompson DR, Obarzanek E, Franko DL, Barton BA, Morrison J, Biro FM, Daniels SR, Striegel-Moore RH. Childhood overweight and cardiovascular disease risk factors: the National Heart, Lung, and Blood Institute Growth and Health Study. J Pediatr. 2007 Jan;150(1):18-25. doi: 10.1016/j.jpeds.2006.09.039. PMID 17188606
- [Background] Hingle MD, O'Connor TM, Dave JM, Baranowski T. Parental involvement in interventions to improve child dietary intake: a systematic review. Prev Med. 2010 Aug;51(2):103-11. doi: 10.1016/j.ypmed.2010.04.014. Epub 2010 May 10. PMID 20462509
- [Derived] Elizondo-Montemayor L, Moreno-Sanchez D, Gutierrez NG, Monsivais-Rodriguez F, Martinez U, Lamadrid-Zertuche AC, Hernandez-Torre MM. Individualized tailor-made dietetic intervention program at schools enhances eating behaviors and dietary habits in obese Hispanic children of low socioeconomic status. ScientificWorldJournal. 2014 Jan 30;2014:484905. doi: 10.1155/2014/484905. eCollection 2014. PMID 24592170